CLINICAL TRIAL: NCT03774732
Title: PD-1 Inhibitor and Chemotherapy With Concurrent Irradiation at Varied Tumour Sites in Advanced Non-small Cell Lung Cancer
Acronym: NIRVANA-LUNG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0107/1718
Record Dates: First submitted 2018-09-26; First posted 2018-12-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; Non-Small Cell Carcinoma of Lung, TNM Stage 4
Keywords: NSCLC; radiotherapy; immunotherapy; PD(L)-1 blockage
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Radiotherapy, Conformal; Radiosurgery; pembrolizumab; Drug Therapy; Carboplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pembrolizumab+ Chemotherapy + Radiotherapy (Experimental): In the experimental arm, patients will receive the same treatment as the control arm (chemotherapy plus pembrolizumab) in addition with conformal 3D radiotherapy (3D-CRT) or stereotactic ablative radiotherapy (SABR) that will be delivered at C2D1, 21 days after the beginning of pembrolizumab using photons/electrons with standard field encompassing tumour.
  Irradiation technique (3D-CRT or SABR) will be at physician discretion. Ideally, oligometastatic patient (defined by the presence of less than 6 metastases) should be treated with SABR and those with non-oligometastatic disease should be treated with 3D-CRT.
  Radiotherapy will be delivered a dose of at least 18 Gy in 3 X 6 Gy for 3D-CRT (cf. protocol for possible schemes and volumes restriction).
  Irradiated tumor size will be ≤5 cm (GTV <65 mL sphere); partial tumor irradiation should be delivered if larger tumor size while respecting dose constraints.
  Interventions: Radiation: Radiotherapy; Drug: Pembrolizumab; Drug: Chemotherapy
- Pembrolizumab+ Chemotherapy (Active Comparator): Squamous-cell lung carcinoma:
  Pembrolizumab every 3 weeks and carboplatin + paclitaxel or nab paclitaxel every 3 weeks for 4 cycles then pembrolizumab every 3 or 6 weeks (according to the current version of the SmPC )
  Non squamous-cell lung carcinoma:
  Pembrolizumab every 3 weeks and carboplatin or cisplatin + pemetrexed every 3 weeks for 4 cycles, and then pemetrexed plus pembrolizumab every 3 weeks (according to the current version of the SmPC)
  Pembrolizumab treatment may be continued as long as patient is experiencing clinical benefit, as assessed by an investigator, in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression after an integrated assessment of radiographic data, biopsy results (if available) and clinical status.
  Interventions: Drug: Pembrolizumab; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Irradiation technique (3D-CRT or SABR) will be at physician discretion.
  Other Names: 3D-CRT or SABR
  Arms: Pembrolizumab+ Chemotherapy + Radiotherapy
Drug: Pembrolizumab — pembrolizumab will be administered as per standard of care every 3 weeks until progression or toxicity
Drug: Chemotherapy — for squamous NSCLC carboplatin AUC6, paclitaxel 200 mg/m² every 3 weeks for 4 cycles; for non-squamous NSCLC carboplatin AUC5 or cisplatin 75 mg/m² every 3 weeks for 4 cycles, and pemetrexed 500 mg/m² every 3 weeks until progression or toxicity
  Other Names: Carboplatin, paclitaxel, nab-paclitaxel, cisplatin, pemetrexed

SUMMARY:
Overall survival (OS) of patients with advanced (stage IIIB/IV) non-small-cell lung cancer (NSCLC) remains short after the first line of treatment with a median OS of 12.2 months in non squamous NSCLC and 9.2 months in squamous NSCLC . In this setting the programmed death 1/ligand 1 (PD-1/-L1) were targeted with nivolumab (IgG4) in advanced squamous and nonsquamous NSCLC leading to an increase of the 1-year OS rate of approximately 10-15% in both histologies. Nivolumab, pembrolizumab and atezolizumab are now considered a standard of care in 2nd line advanced NSCLC and in 1st line for pembrolizumab but but prognosis still remains poor in advanced NSCLC. Overall survival (OS) of patients with advanced (stage III/IV) NSCLC remains limited with a median OS of 12.2 months in non-squamous NSCLC and 9.2 months in squamous NSCLC if anti-PD1 alone. It is of around 16 months if pembrolizumab is combined with chemotherapy.

Preclinical data indicates that anti-tumor efficacy is increased when anti-PD-1/-L1 are combined with irradiation (IR). Radiotherapy alone can elicit tumor cell death which can increase tumor antigen in the blood stream, favoring recognition by the immune system and its activation against tumor cells outside of the radiation field (="abscopal effect").

IR may also reverse acquired resistance to PD-1 blockade immunotherapy by limiting T-cell exhaustion.

Because of these preclinical and clinical data several studies analysing the combination of IR and anti-PD1 in NSCLC are ongoing. Among them, two studies are testing the administration of IR and nivolumab in stage III NSCLC: the NCT02768558 phase III trial (RTOG), and the NCT02434081 phase II trial (ETOP). Antonia et al [2017] tested the use of anti-PD-L1 after chemoradiotherapy in unresectable stage III NSCLC. Median time to distant metastasis was increased (23.2 months vs. 14.6 months, p<0.001). An increase of OS is consequently expected.

However, no study involving concurrent RT and pembrolizumab combined with chemotherapy in advanced NSCLC is ongoing, which is the purpose of the present study, NIRVANA-Lung.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Patient must have signed a written informed consent form prior to any study specific procedures
2. Histologically or cytologically confirmed advanced (stage IIIB/IIIC/IV), squamous or non-squamous NSCLC
3. NSCLC patients eligible for treatment with pembrolizumab and chemotherapy according to the European Marketing Authorization:

   1. squamous: in combination with carboplatin and either paclitaxel or nab-paclitaxel
   2. non squamous with no EGFR or ALK positive mutations: in combination with pemetrexed and a platinum based chemotherapy
4. Patient ≥18 of age
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
6. Life expectancy >3 months
7. Measurable lesion as assessed by RECIST version 1.1
8. Metastases and/or primary tumour eligible for 3 dimensional conventional radiotherapy (3D-CRT) or stereotactic ablative radiotherapy (SABR) in terms of dose constraints at organ at risk (according to QUANTEC review)
9. Patients must have adequate organ function defined by the following laboratory results obtained within 14 days prior to the first study treatment:

   1. absolute neutrophil count of ≥1 500 /mm³
   2. platelets ≥ 100 000/mm³
   3. haemoglobin >9 g/dL (transfusions allowed)
   4. creatinine clearance >60 mL/min
   5. bilirubin ≤1.5 X upper limit of normal (ULN) (unless Gilbert's syndrome where 3 X ULN is permitted)
   6. serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 X ULN (unless documented liver metastasis where ≤5 X ULN is permitted)
   7. Alkaline phosphatase (ALP) ≤2.5 X ULN (unless documented bone or liver metastasis where ≤5 X ULN is permitted)
   8. International normalized ratio (INR), prothrombin (PT), and prothrombin time (PTT) ≤1.5 X ULN (unless the subject is receiving anticoagulant therapy)
10. Woman of childbearing potential and male patients must agree to use adequate contraception for the duration of study participation and up to 6 months after completing treatment/therapy
11. Patients affiliated to the social security system (or equivalent)
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits, and examinations including follow-up

NON-INCLUSION CRITERIA:

1. Non-squamous NSCLC with targetable tumor mutations, activating EGFR mutations or ALK translocation Note: documentation of these mutation for non-squamous histology is mandatory as standard of care
2. Stage IIIB/IIIC NSCLC patient eligible to curative (thoracic radiotherapy or surgery) treatments in first line treatment
3. Prior therapy with T-cell costimulation or checkpoint-targeted agents Note: Stage I-III NSCLC who previously received single-agent anti-PD(L)1 immunotherapy and ultimately develop metastases remain eligible (minimal immunotherapy washout period of 3 months)
4. Clinical need of radiotherapy (e.g.: whole brain irradiation, painful metastasis, bleeding, compressive metastases)
5. Irradiation within 2 months before inclusion
6. Leptomeningeal carcinomatosis, or metastases with indistinct borders making targeting not feasible
7. Patient with evidence of active (presence of symptoms or requiring steroid treatment) central nervous system (CNS) metastases and/or carcinomatous meningitis. Patient with brain metastasis can be included if asymptomatic and not requiring steroids
8. Metastases located within 3 cm of the previously irradiated structures (EQD2doses):

   1. Spinal cord previously irradiated to >40 Gy;
   2. Brachial plexus previously irradiated to >50 Gy;
   3. Small intestine, large intestine, or stomach previously irradiated to >45 Gy;
   4. Brainstem previously irradiated to >50 Gy;
   5. Lung previously irradiated with prior V20Gy >30%
9. Active autoimmune disease except vitiligo, type-1 diabetes, hypothyroid stabilized with hormonal substitution, psoriasis
10. Symptomatic interstitial lung disease
11. Systemic immunosuppression or systemic immunosuppressive medicinal products within 2 weeks prior to study entry
12. Concomitant treatment with steroids > 10 mg Note1: higher dose of steroids can be prescribed in case of occurrence of toxicities during radiotherapy; prophylactic dose of maximum 1 mg per kg during 2 weeks are authorized during the delivery of more than 6 Gy per fraction Note2: temporary use of steroid (less than 4 weeks) at a dose of 1 mg/kg is accepted
13. Prior invasive malignancy within the past 2 years (except non-melanomatous skin cancer non-invasive carcinoma in-situ of the breast, oral cavity, bladder or cervix)
14. Known Acquired Immune Deficiency Syndrome (AIDS) or severe uncontrolled co-morbidity
15. Known currently active infection including hepatitis B and hepatitis C
16. Patient who was administered a live, attenuated vaccine within 28 days prior to enrolment
17. Patient with any other disease or illness that requires hospitalisation or is incompatible with the study treatment are not eligible. Patient unable to comply with study obligations for geographic, social, or physical reasons, or who is unable to understand the purpose and procedures of the study
18. Patient who have taken any investigational medicinal product or have used an investigational device within 30 days of inclusion
19. Pregnant or breast feeding woman
20. Person deprived of their liberty or under protective custody or guardianship
21. If pemetrexed: patient is unable or unwilling to take folic acid or vitamin B12 supplementation
22. Pre-existing peripheral neuropathy of a severity of grade ≥ 2 by NCI CTCAE v5.0
23. Known hypersensitivity to one of the compounds or substances used in this protocol
24. Major surgery within the 28 days before initiating study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Estimated)
Dates: Start 2018-01-24 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
1-year Overall Survival | 1 year
  The primary endpoint of this trial is overall survival (OS) defined as the time from randomization to the date of documented death from any cause or last follow-up.

SECONDARY OUTCOMES:
Tumour response | 1 year
  Tumour response is defined as the percentage of patients with a complete response (CR) or partial response (PR), according to RECIST 1.1 and iRECIST (centralized response evaluation).
Progression-free survival | 1 year
  Progression-free survival (PFS) is defined as the time from randomization until documented disease progression (PD) according to RECIST 1.1 and iRECIST (centralized response evaluation for both arms), or death, whichever occurs first.
Local and distant controls in irradiated patients | 6 months and 1 year
  Local and distant controls in irradiated patients are defined as the time from randomization to the first documented local event or distant event.
Quality of life of the patients using EORTC-QLQ-C 30 | up to 2 years
  Quality of life will be assessed using QLQ-C 30 questionnaire from the European Organization for Research and Treatment of Cancer (EORTC). It is a 30-item self-reporting questionnaire developed to assess the quality of life of cancer patients. It is grouped into five functional subscales (role, physical, cognitive, emotional and social functioning). In addition, there are three multi-item symptom scales (fatigue, pain, and nausea and vomiting), individual questions concerning common symptoms in cancer patients,and two questions assessing overall Quality of Life
Acute/Late toxicities | 1 year
  Acute/ late toxicity will be assessed according to the flowchart and graded by CTCAE v5
Non-small lung cancer specific survival | 1 year
  To evaluate, compared to standard of care, whether the addition of radiotherapy improves survival of patients until death from non-small lung cancer
2-year Overall survival | 2 years
  Overall survival (OS) is defined as the time from randomization to the date of documented death from any cause or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DOYEN, MD, Principal Investigator — Centre Antoine Lacassagne; Antonin LEVY, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Benjamin BESSE, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (58):
- France (57):
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Centre Marie Curie, Arras
  - Hôpital Privé Arras Les Bonnettes, Arras
  - Institut Sainte Catherine, Avignon
  - Centre Pierre Curie, Beuvry
  - Clinique Ambroise Pare, Beuvry
  - Hôpital Simone Veil Blois, Blois
  - Institut Bergonie, Bordeaux
  - CHRU de Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier Universitaire De Caen - Hôpital Cote De Nacre, Caen
  - Centre Hospitalier Dr Jean-Eric TECHER, Calais
  - Centre hospitalier de Cannes Simone Veil, Cannes
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Institut de Cancérologie de Bourgogne, Chalon-sur-Saône
  - Pôle départemental de Cancérologie Libérale 37, Chambray-lès-Tours
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal De Creteil, Créteil
  - Centre Georges Francois Leclerc, Dijon
  - Institut de Cancérologie de Bourgogne, Dijon
  - Polyclinique du Parc Drevon, Dijon
  - Centre André DUTREIX, Dunkirk
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Centre de radiothérapie et de cancérologie de Blois, La Chaussée-Saint-Victor
  - CHU Sud de la Réunion, La Réunion
  - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Centre Oscar Lambret, Lille
  - Clinique Chenieux, Limoges
  - Hôpital Européen Marseille, Marseille
  - Hôpital Privé Clairval, Marseille
  - Centre Hospitalier de Montelimar, Montélimar
  - Centre de cancérologie du grand Montpellier-Clinique Clementville, Montpellier
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - Centre Azuréen De Cancérologie, Mougins
  - Hôpital Privé Arnault Tzanck, Mougins
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Fondation Hôpital Saint-Joseph, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Tenon, Paris
  - Centre Catalan d'Oncologie, Perpignan
  - Institut Jean Godinot, Reims
  - Centre Frédéric JOLIOT, Rouen
  - Centre Henri Becquerel, Rouen
  - Clinique Saint-Hilaire, Rouen
  - Hopital Charles Nicolle, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - CHU St Etienne, Saint-Etienne
  - Centre Joliot Curie, Saint-Martin-Boulogne
  - Centre Paul Strauss, Strasbourg
  - Polyclinique de l'Ormeau, Tarbes
  - CHU de Toulouse Hôpital Larrey, Toulouse
  - Institut Claudius Regaud, Toulouse
  - Centre Marie Curie, Valence
  - Hôpital Privé Drôme Ardèche, Valence
  - Institut De Cancerologie De Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Centre Hospitalier Princesse Grace, Monaco, Monaco

REFERENCES:
- [Derived] Doyen J, Besse B, Texier M, Bonnet N, Levy A. PD-1 iNhibitor and chemotherapy with concurrent IRradiation at VAried tumor sites in advanced Non-small cell lung cAncer: the Prospective Randomized Phase 3 NIRVANA-Lung Trial. Clin Lung Cancer. 2022 May;23(3):e252-e256. doi: 10.1016/j.cllc.2021.10.008. Epub 2021 Oct 24. PMID 34810130